CLINICAL TRIAL: NCT05922969
Title: Safety of Low PEEP Maneuvers During ARDS Management
Acronym: DEBAS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier VALENCIENNES (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0165
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome; Positive End Expiratory Pressure
Keywords: Acute Respiratory distress syndrome; Positive end expiratory pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute Respiratory distress syndrome (ARDS) is a severe condition in which protective ventilation is a critical point in its management. Positive end expiratory pressure (PEEP) setting can be challenging for clinicians and high PEEP has been associated with better outcome in moderate and severe ARDS. Recently, recruitment to inflation ratio and airway closure have been investigated in order to help PEEP adjustment. However, ventilatory maneuvers are performed with a low level of PEEP and therefore expose to derecruitment and oxygen desaturation. So far, the risk of oxygen desaturation has not been investigated and risk factors are unknown.

The aim of this study is to evaluate the prevalence of oxygen desaturation during ventilatory maneuvers at low level of PEEP in patients with moderate or severe ARDS

ELIGIBILITY:
Inclusion Criteria:

* age : > 18 yo
* inclusion criteria: ARDS, Mechanical ventilation, low PEEP maneuvers

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PEEP in patients with moderate or severe ARDS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-28 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
prevalence of oxygen desaturation | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No